CLINICAL TRIAL: NCT05108610
Title: Shi-style Cervical Manipulations for Nonspecific Neck Pain: a Multi-center, Randomized, Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Beijing Hospital (Other Government); Shenzhen Pingle Orthopaedic Hospital (Unknown); Dongzhimen Hospital, Beijing (Other); Traditional Chinese Medicine Hospital of the Ningxia Hui Autonomous Region (Other); Traditional Chinese Medicine Hospital of Ganzhou Nankang District (Unknown)
Responsible Party: Principal Investigator, Cui xuejun, Clinical Research Base of Traditional Chinese Medicine, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Nonspecific Neck Pain
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Nonspecific Neck Pain
Keywords: Randomized controlled study；nonspecific neck pain；Shi-style manipulations；Mechanical parameters

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traction (Active Comparator): 6kg to 10kg, 3 times a week, once the other day（except the weekends）,20 minutes, 2 weeks.
  Interventions: Other: Cervical Traction control
- Shi-style manipulations (Experimental): Shi-style manipulations is a cervical manipulation for cervical spondylosis.This manipulation is a kind of traditional Chinese massage and it can dredge the meridians. Patients are treated every day for 30 minutes. Seven times as one course and totally there are two courses. 3 times a week, once the other day（except the weekends）,30 minutes, 2 weeks.
  Interventions: Other: Shi-style manipulations

INTERVENTIONS:
Other: Shi-style manipulations — Shi-style cervical manipulation is a spinal manipulation for cervical radiculopathy.It is a kind of traditional chinese massage and can dredge the meridian.Patients are treated every day for 30 minutes.Seven times at one course and totally there are two courses.3 times a week, once the other day（except the weekends）,30 minutes, 2 weeks.
  Other Names: manipulations for cervical radiculopathy
  Arms: Shi-style manipulations
Other: Cervical Traction control — 6kg to 10kg, 3 times a week, once the other day（except the weekends）,20 minutes, 2 weeks.
  Other Names: Cervical traction
  Arms: Traction

SUMMARY:
Spinal instability diseases have a high prevalence and great harm. The research on how to prevent and treat degenerative spinal instability diseases has become a hot spot in the international academic community, and it is also an important research content in the field of "population and health" in my country. Clinical studies have shown that the "Shi-style manipulations" have outstanding efficacy and high safety in the treatment of degenerative spinal instability diseases. The study intends to carry out a randomized, traction-controlled study in 5 tertiary hospital test centers, with patients with non-specific neck pain as the research object, using "Shi-style manipulations" and traction as intervention methods, and checking indicators and subjective effects through relevant instruments Indicators, quantitative verification of the mechanical parameters and biological effects of the "Shi-style manipulations", scientific evaluation of the efficacy and safety of the "Shi-style manipulations" in non-specific neck pain diseases.

DETAILED DESCRIPTION:
Spinal diseases are listed as the second most serious diseases in the world's top ten Diseases released by WHO. With the rapid pace of life, the aging of the population and the increase in chronic strain, the incidence of degenerative spinal instability diseases remains high and medical expenses increase.

From 1999 to 2006, 534 patients with various types of degenerative spine instability diseases (except myelomyelitis) were treated by the project team, and the total effective rate of the "three steps and nine steps" in the treatment of clinical symptoms and signs of degenerative spine instability diseases was 91.76%. Through reviewing 60 cases of nerve root type of randomized controlled trials, 8 weeks after treatment, treatment group 30 cases (the whole neck three-step nine method), total effective rate 93.3%, control group total effective rate was 73.3% (cervical traction) (P < 0.01), the treatment group in improving the neck shoulder pain, upper limb numbness, dizziness, tinnitus, brachial plexus pull test is better than that in control group (P < 0.05), the clinical operation without adverse reaction.

Clinical studies have shown that the "Shi-style manipulations" have outstanding efficacy and high safety in the treatment of degenerative spinal instability diseases. The study intends to carry out a randomized, traction-controlled study in 5 tertiary hospital test centers, with patients with non-specific neck pain as the research object, using "Shi-style manipulations" and traction as intervention methods, and checking indicators and subjective effects through relevant instruments Indicators, quantitative verification of the mechanical parameters and biological effects of the "Shi-style manipulations", scientific evaluation of the efficacy and safety of the "Shi-style manipulations" in non-specific neck pain diseases.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis is non-specific neck pain;
* Male or female between the ages of 18 and 65 (including 18 and 65);
* VAS score ≥30 mm;
* Sign the informed consent voluntarily.

Exclusion Criteria:

* Have received surgical treatment or neck trauma for cervical spondylosis in the past;
* With cervical nerve compression or spinal cord compression symptoms and signs, MRI found spinal compression;
* The vertebral body was shifted, horizontally shifted >3 mm forward, backward or laterally, and the adjacent intervertebral space had an Angle difference of >11°;
* Patients with liver, kidney, hematopoietic system and other serious primary diseases, with a history of opioid analgesics, sedative and hypnotic drugs and alcohol abuse;
* Patients with osteoporosis, spinal tuberculosis, vertebral body malformation, malignant tumors and mental diseases;
* Pregnant women and lactating women;
* Unable to participate in the follow-up (for example, the plan of migration or long-distance relocation within half a year, no communication tools such as mobile phones, etc.), and the patients without the ability to participate in the half-year follow-up cannot read and write Chinese;
* received radio frequency, minimally invasive, ozone, small needle knife, manipulation, traction or closed treatment Within the last two weeks;
* Participating in other clinical trials related to cervical spondylosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal ultrasound | changes from baseline at 2 weeks
  Measure the ratio of the muscle thickness of the back of the neck muscles to the strain rate of the back of the neck muscles.Use real-time dual-frame imaging to adjust the area of interest to ensure coverage of trapezius, supraspinatus, infraspinatus, levator scapula, and sternocleidomastoid. During operation, the probe lightly touches the ultrasonic coupling patch and is perpendicular to the body surface, hold the probe to slightly vibrate up and down, and keep the pressure release index at 3-4. Collect the elastic image to ensure that the image is clear and stable for 3-4 seconds. Observe the elastic image and outline the reference area and the area of interest. Calculate the SR values of the reference area and the area of interest with the software that comes with the ultrasound system. Measure 3 times and take the average value.
Visual Analogue scale，(VAS) | changes from baseline at 2 weeks
  The visual analog scale is used to measure the patient's current pain level.This scoring ruler has a scale in centimeters on one side, and the smallest scale is millimeters; on the other side, the two ends are marked as "painless" and "most painful". When using, the researcher holds both ends of the visual analog scale with both hands. The scale faces the researcher and the non-scale faces the patient. The patient is asked to use the thumb and index finger to move the upper scale of the ruler to the level of pain.Read the scale value corresponding to the red line of the vernier of the visual analog scale and record it in the research medical record. The value is rounded to a single digit, and the unit is millimeter (mm). The red line is between the two scales, and the left value is taken. Such as "53mm".
pressure pain threshold | changes from baseline at 2 weeks
  Determine the corresponding acupoints on the subject's neck, use a round probe to find the pain sensitive points, and mark them with a marker to be measured. There are 10 points in total.In order to fully relax the tested muscles, supine or lateral positions are used in the measurement. Before measuring, inform the subject of the entire operation process.The measurement was started after he entered the examination room and rested quietly for 5 minutes. During the measurement, a tester holds a digital dynamometer, touches the instrument probe vertically downwards to the skin, and applies pressure to the test point at a uniform speed when applying force. When the subject begins to feel pain, immediately remove the test probe and read the data on the instrument at the same time. After the measurement is completed, press the zero button to perform the next measurement. The same acupuncture point was tested 3 times with an interval of 30s, and the average value was taken.
Musculoskeletal ultrasound | changes from baseline at 1 month
  Measure the ratio of the muscle thickness of the back of the neck muscles to the strain rate of the back of the neck muscles.Use real-time dual-frame imaging to adjust the area of interest to ensure coverage of trapezius, supraspinatus, infraspinatus, levator scapula, and sternocleidomastoid. During operation, the probe lightly touches the ultrasonic coupling patch and is perpendicular to the body surface, hold the probe to slightly vibrate up and down, and keep the pressure release index at 3-4. Collect the elastic image to ensure that the image is clear and stable for 3-4 seconds. Observe the elastic image and outline the reference area and the area of interest. Calculate the SR values of the reference area and the area of interest with the software that comes with the ultrasound system. Measure 3 times and take the average value.
Visual Analogue scale，(VAS) | changes from baseline at 1 month
  The visual analog scale is used to measure the patient's current pain level.This scoring ruler has a scale in centimeters on one side, and the smallest scale is millimeters; on the other side, the two ends are marked as "painless" and "most painful". When using, the researcher holds both ends of the visual analog scale with both hands. The scale faces the researcher and the non-scale faces the patient. The patient is asked to use the thumb and index finger to move the upper scale of the ruler to the level of pain.Read the scale value corresponding to the red line of the vernier of the visual analog scale and record it in the research medical record. The value is rounded to a single digit, and the unit is millimeter (mm). The red line is between the two scales, and the left value is taken. Such as "53mm".
pressure pain threshold | changes from baseline at 1 month
  Determine the corresponding acupoints on the subject's neck, use a round probe to find the pain sensitive points, and mark them with a marker to be measured. There are 10 points in total.In order to fully relax the tested muscles, supine or lateral positions are used in the measurement. Before measuring, inform the subject of the entire operation process.The measurement was started after he entered the examination room and rested quietly for 5 minutes. During the measurement, a tester holds a digital dynamometer, touches the instrument probe vertically downwards to the skin, and applies pressure to the test point at a uniform speed when applying force. When the subject begins to feel pain, immediately remove the test probe and read the data on the instrument at the same time. After the measurement is completed, press the zero button to perform the next measurement. The same acupuncture point was tested 3 times with an interval of 30s, and the average value was taken.
Musculoskeletal ultrasound | changes from baseline at 3 months
  Measure the ratio of the muscle thickness of the back of the neck muscles to the strain rate of the back of the neck muscles.Use real-time dual-frame imaging to adjust the area of interest to ensure coverage of trapezius, supraspinatus, infraspinatus, levator scapula, and sternocleidomastoid. During operation, the probe lightly touches the ultrasonic coupling patch and is perpendicular to the body surface, hold the probe to slightly vibrate up and down, and keep the pressure release index at 3-4. Collect the elastic image to ensure that the image is clear and stable for 3-4 seconds. Observe the elastic image and outline the reference area and the area of interest. Calculate the SR values of the reference area and the area of interest with the software that comes with the ultrasound system. Measure 3 times and take the average value.
Visual Analogue scale，(VAS) | changes from baseline at 3 months
  The visual analog scale is used to measure the patient's current pain level.This scoring ruler has a scale in centimeters on one side, and the smallest scale is millimeters; on the other side, the two ends are marked as "painless" and "most painful". When using, the researcher holds both ends of the visual analog scale with both hands. The scale faces the researcher and the non-scale faces the patient. The patient is asked to use the thumb and index finger to move the upper scale of the ruler to the level of pain.Read the scale value corresponding to the red line of the vernier of the visual analog scale and record it in the research medical record. The value is rounded to a single digit, and the unit is millimeter (mm). The red line is between the two scales, and the left value is taken. Such as "53mm".
pressure pain threshold | changes from baseline at 3 months
  Determine the corresponding acupoints on the subject's neck, use a round probe to find the pain sensitive points, and mark them with a marker to be measured. There are 10 points in total.In order to fully relax the tested muscles, supine or lateral positions are used in the measurement. Before measuring, inform the subject of the entire operation process.The measurement was started after he entered the examination room and rested quietly for 5 minutes. During the measurement, a tester holds a digital dynamometer, touches the instrument probe vertically downwards to the skin, and applies pressure to the test point at a uniform speed when applying force. When the subject begins to feel pain, immediately remove the test probe and read the data on the instrument at the same time. After the measurement is completed, press the zero button to perform the next measurement. The same acupuncture point was tested 3 times with an interval of 30s, and the average value was taken.

SECONDARY OUTCOMES:
Neck Disabilitv Index， (NDI) | changes from baseline at 2 weeks
  The Neck Disability Index (NDI) is one of the most frequently used questionnaires in clinical practice. The questionnaire mainly assesses the patient's pain level, self-care ability, weightlifting, reading, headache level, concentration, work, driving, sleep, and entertainment. It quantifies the points of all aspects, and the score ranges from 0 points (no disability) to 5 points (completely disabled), the total score ranges from 0 points (no disability) to 50 points (completely disabled), for a total of 50 points. The lower the total score, the less severe the patient's condition, and vice versa.
the MOS item short from health survey，(SF-36) | changes from baseline at 2 weeks
  The SF-36 scale is a universal scale developed by the American Medical Research Group to measure the quality of life, and is universally recognized and widely used in the world. This scale has a total of 8 dimensions to evaluate health-related quality of life (HRQOL), which is divided into two categories: physical health and mental health, namely physical function (PF), physical function (RP), physical pain (BP), and general health (CH), Activity (VT), Social Function (SF), Emotional Function (RE), Mental Health (MH).
Cervical range of motion | changes from baseline at 2 weeks
  Measure the range of cervical spine flexion, extension, lateral flexion, and rotation by using a universal protractor
Neck Disabilitv Index， (NDI) | changes from baseline at 1 month
  The Neck Disability Index (NDI) is one of the most frequently used questionnaires in clinical practice. The questionnaire mainly assesses the patient's pain level, self-care ability, weightlifting, reading, headache level, concentration, work, driving, sleep, and entertainment. It quantifies the points of all aspects, and the score ranges from 0 points (no disability) to 5 points (completely disabled), the total score ranges from 0 points (no disability) to 50 points (completely disabled), for a total of 50 points. The lower the total score, the less severe the patient's condition, and vice versa.
the MOS item short from health survey，(SF-36) | changes from baseline at 1 month
  The SF-36 scale is a universal scale developed by the American Medical Research Group to measure the quality of life, and is universally recognized and widely used in the world. This scale has a total of 8 dimensions to evaluate health-related quality of life (HRQOL), which is divided into two categories: physical health and mental health, namely physical function (PF), physical function (RP), physical pain (BP), and general health (CH), Activity (VT), Social Function (SF), Emotional Function (RE), Mental Health (MH).
Cervical range of motion | changes from baseline at 1 month
  Measure the range of cervical spine flexion, extension, lateral flexion, and rotation by using a universal protractor
Neck Disabilitv Index， (NDI) | changes from baseline at 3 months
  The Neck Disability Index (NDI) is one of the most frequently used questionnaires in clinical practice. The questionnaire mainly assesses the patient's pain level, self-care ability, weightlifting, reading, headache level, concentration, work, driving, sleep, and entertainment. It quantifies the points of all aspects, and the score ranges from 0 points (no disability) to 5 points (completely disabled), the total score ranges from 0 points (no disability) to 50 points (completely disabled), for a total of 50 points. The lower the total score, the less severe the patient's condition, and vice versa.
the MOS item short from health survey，(SF-36) | changes from baseline at 3 months
  The SF-36 scale is a universal scale developed by the American Medical Research Group to measure the quality of life, and is universally recognized and widely used in the world. This scale has a total of 8 dimensions to evaluate health-related quality of life (HRQOL), which is divided into two categories: physical health and mental health, namely physical function (PF), physical function (RP), physical pain (BP), and general health (CH), Activity (VT), Social Function (SF), Emotional Function (RE), Mental Health (MH).
Cervical range of motion | changes from baseline at 3 months
  Measure the range of cervical spine flexion, extension, lateral flexion, and rotation by using a universal protractor

OTHER OUTCOMES:
The doctor of traditional Chinese medicine syndrome | changes from baseline at 2 weeks
  The TCM Syndrome Feature Scale is based on the patient's general symptoms, signs (including tongue and pulse), physical examination, and laboratory examination results to establish an information table, and then use the difference matrix method to perform attribute reduction and case reduction to obtain The lower approximation set and the upper approximation set are used to extract the definite rules and possible rules of TCM diagnosis. In this way, the subjectivity and one-sidedness of doctors are avoided to a large extent, making TCM syndrome diagnosis and treatment more standardized and scientific
The doctor of traditional Chinese medicine syndrome | changes from baseline at 1 month
  The TCM Syndrome Feature Scale is based on the patient's general symptoms, signs (including tongue and pulse), physical examination, and laboratory examination results to establish an information table, and then use the difference matrix method to perform attribute reduction and case reduction to obtain The lower approximation set and the upper approximation set are used to extract the definite rules and possible rules of TCM diagnosis. In this way, the subjectivity and one-sidedness of doctors are avoided to a large extent, making TCM syndrome diagnosis and treatment more standardized and scientific
The doctor of traditional Chinese medicine syndrome | changes from baseline at 3 months
  The TCM Syndrome Feature Scale is based on the patient's general symptoms, signs (including tongue and pulse), physical examination, and laboratory examination results to establish an information table, and then use the difference matrix method to perform attribute reduction and case reduction to obtain The lower approximation set and the upper approximation set are used to extract the definite rules and possible rules of TCM diagnosis. In this way, the subjectivity and one-sidedness of doctors are avoided to a large extent, making TCM syndrome diagnosis and treatment more standardized and scientific

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wan, Doctor of Medicine(M.D.), Principal Investigator — Shanghai University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No